CLINICAL TRIAL: NCT05396794
Title: Bariatric Surgery Among Women With Obesity and Low Risk Endometrial Cancer: A Pilot Study
Brief Title: Bariatric Education for Women With Obesity and Endometrial Cancer
Acronym: SCC-BAREDU
Status: Terminated | Type: Observational
Why Stopped: No Surgeon to perform the operations.
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Other Study IDs: OU-SCC-BAREDU
Record Dates: First submitted 2022-05-11; First posted 2022-05-31 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Obesity; Endometrial Cancer; Bariatric Surgery Candidate
Keywords: bariatric surgery; endometrial cancer; obesity
MeSH Terms: conditions — Obesity; Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control Group: If the patient is in group 1, she will get standard education for weight loss, which will be provided by her Gynecologic Oncologist. This will take about 15 minutes.
  Interventions: Behavioral: Standard weight loss education
- Video Group: If the patient is in group 2, she will get standard education for weight loss provided by her Gynecologic Oncologist. Then she will be asked to view a 15-minute video to get information regarding obesity, the relationship of obesity and endometrial cancer, and the safety and benefits of bariatric surgery. These will take about 30 minutes.
  Interventions: Behavioral: Standard weight loss education + Educational Video

INTERVENTIONS:
Behavioral: Standard weight loss education — Participants will be randomized and given the standard weight loss education by the Gynecologic Oncology provider.
  Groups: Control Group
Behavioral: Standard weight loss education + Educational Video — Participants will be randomized and given the standard weight loss education by the Gynecologic Oncology provider followed by a 15-minute educational video detailing the benefits of weight loss.
  Groups: Video Group

SUMMARY:
The purpose of this study is to examine whether a standardized video education tool will improve knowledge regarding obesity and bariatric surgery and increase bariatric surgery referrals for obese women with endometrial cancer.

DETAILED DESCRIPTION:
An estimated 50% of all endometrial cancer cases are associated with obesity. Bariatric surgery has been shown to reduce the risk of hormone-related cancers, including endometrial cancer, by up to 70-80%. This prospective, study of 80 patients will be randomized to either a standard education for weight loss provided by their oncologist or a standard education plus a 15-minute video with information regarding obesity, relationship of obesity and endometrial cancer, and the safety and benefits of bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-80 with class II or greater obesity (BMI ≥ 35)
* Have pathologically-confirmed endometrial cancer
* Have completed initial therapy (e.g. surgery, hormonal therapy, vaginal cuff brachytherapy, or a combination of these modalities) and require no further interventions related to cancer care. Patients taking hormonal therapy as part of cancer treatment may be included.

Exclusion Criteria:

* Under the age of 18 or over the age of 80
* Have previously undergone bariatric surgery
* Requires ongoing cancer treatment with chemotherapy or whole pelvic radiation.
* Poor surgical candidate secondary to comorbidities or performance status.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This study will include women only as it is focused on a sex-specific cancer (endometrial).
Study Population: Women with endometrial cancer with obesity who are receiving care at the Stephenson Cancer Center will be considered for inclusion. All patients regardless of race, ethnicity, or socioeconomic status will be included without discrimination.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
Proportion of patient's obesity relevant knowledge pre- and post-education intervention | 6 Months
  Proportion of patient will complete a pre and post (6 months after enrollment) survey to examine the knowledge of obesity, endometrial cancer and bariatric surgery. These measures will be self-reported 6 months after the patient was educated on the benefits of weight loss.
Proportion of patients who chose to take part in bariatric surgery. | 6 Months
  Based on these pre-and post-educational surveys patient's decision to participate or to decline the bariatric surgery referral will be recorded, including the patients experience with bariatric surgery program.

CONTACTS AND LOCATIONS:
Overall Officials: Laura L Holman, MD, Principal Investigator — University of Oklahoma Stephenson Cancer Center
Locations (1):
- Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No